CLINICAL TRIAL: NCT00300729
Title: Cox-2-Inhibitor and Chemotherapy in Non-Small Cell Lung Cancer. A Prospective Randomized Double-Blind Study
Brief Title: Effect of Celecoxib on Survival in Patients With Advanced Non-Small Cell Lung Cancer Receiving Chemotherapy
Acronym: CYCLUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Swedish Lung Cancer Study Group (Network); Pfizer (Industry)
Responsible Party: Sverre Sörenson, MD, PhD, Swedish Lung Cancer Study Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLCSG0501
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Cyclooxygenase-2 inhibitors; Celecoxib; Carcinoma, non-small-cell lung; Antineoplastic agents; Therapy, palliative; Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Active Comparator): Four cycles of combination chemotherapy, usually with carboplatin + gemcitabine or carboplatin + vinorelbine, plus celecoxib 400 mg b.i.d. Treatment with celecoxib is continued after completion of chemotherapy. Maximum treatment duration is one year.
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Chemotherapy as in arm 1 plus placebo capsules, b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 400 mg twice daily, orally, starting on the same day as palliative chemotherapy. Maximum duration of treatment is one year. Treatment should be terminated earlier in case of disease progression, unacceptable toxicity, or if the patient wants to stop treatment.
  Other Names: Celebra; Onsenal
  Arms: Celecoxib
Drug: Placebo — One capsule twice daily, starting on the same day as palliative chemotherapy. Maximum duration of treatment is one year. Treatment should be terminated earlier in case of disease progression, unacceptable toxicity, or if the patient wants to stop treatment.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to investigate if daily treatment with celecoxib, an inhibitor of cyclooxygenase-2, can prolong survival in patients with advanced non-small cell lung cancer who receive anticancer chemotherapy as their primary treatment. Secondary endpoints of the study are: health-related quality of life, toxicity, cardiovascular events, progression-free survival, and biological markers (VEGF, proteomics).

DETAILED DESCRIPTION:
The study (CYCLUS trial, CY-cyclooxygenase-2 inhibitor, Chemotherapy, LUng cancer, Survival) is a prospective randomized double-blind multicenter trial. Patients are randomized to receive celecoxib at a dose of 400 mg b.i.d. or placebo. Primary endpoint of the trial is survival. Secondary endpoints are: quality of life, progression-free survival, toxicity, cardiovascular events, and biological parameters (plasma VEGF and proteomics).

The rationale behind the study consists of preclinical observations of antitumor effect of celecoxib in NSCLC. Inhibition of angiogenesis and proliferation as well as increased apoptosis has been demonstrated. In addition, pilot studies have shown that the combination of chemotherapy and celecoxib is feasible. No unexpected toxicity has been recorded in such trials. Furthermore, a randomized study of indomethacin, prednisolone or placebo in other types of advanced cancer, mainly gastrointestinal, showed a survival advantage for patients receiving antiinflammatory treatment.

Chemotherapy is given according to the current standard of the participating institution. In practice, patients will usually receive either carboplatin + gemcitabine or carboplatin + vinorelbine. Treatment duration with chemotherapy is 4 cycles (cycle length 3 weeks) in the absence of tumour progression or prohibitive toxicity.

Treatment with the study drug starts on the first day of cancer chemotherapy. Maximum treatment duration is one year. Treatment will be stopped earlier in case of objective tumor progression, serious toxicity that is considered to be related to the study drug or if the patient wants to stop treatment.

The size of the study is based on the hypothesis that celecoxib could prolong median survival by 8 weeks as compared to 7.5 months in the placebo group. With standard statistical requirements (type I error 5%, type II error 20%), the calculated number of patients was 760.

The study was supported by the Swedish Lung Cancer Study Group and organized as a multicenter trial, with participation of seven university hospitals and six smaller hospitals. The number of new cases of NSCLC stage IIIB-IV and performance status 0-2 in Sweden is around 1200/year. It was expected that 20% of the patients could be included in the study, which would make completion possible in three years.

The study was opened for randomization on May 31, 2006. Recruitment of patients was lower than expected. The study was closed for further randomization on May 31, 2009, as originally planned. 319 patients were included. Since maximum duration of treatment with the study drug is one year, the code will be broken after May 31, 2010. Data analysis is planned to take place in summer and autumn, 2010.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC).
* Age at least 18 years. No upper age limit.
* Disease stage IIIB or IV.
* Performance status (WHO) 0-2
* Treatment with curative intent is not possible
* No prior chemotherapy for the present disease
* Planned treatment is palliative chemotherapy
* WBC count at least 3.0, platelet count at least 100
* Bilirubin < 1.5 * upper reference limit (URL), ASAT and ALAT < 3 * URL (<5 in case of liver metastases)
* Calculated creatinine clearance at least 40 mg/ml
* Informed oral and written consent

Exclusion criteria:

* Regular use of NSAID (except ASA at a dose of 50-100 mg daily)
* Active duodenal ulcer, ongoing gastrointestinal bleeding or inflammatory bowel disease
* Serious heart failure or serious liver disease
* Hypersensitivity so sulfonamides
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Minimum follow-up 1 yr after randomization

SECONDARY OUTCOMES:
Quality of life | Week 0, 3, 6, 9, 12, 20, 28, 36, 44
Progression-free survival | minimum follow-up 1 yr after randomization
Toxicity | Within one month after stopping study drug
Cardiovascular events | Within one month after stopping study drug
Biological parameters (plasma VEGF, proteomics) | Week 0, 6, 12, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Sörenson, MD, PhD, Study Chair — Department of Medicine, Ryhov County Hospital, Jönköping, Sweden, Department of Pulmonary Medicine, University Hospital, Linköping, Sweden, and Department of Medical and Health Sciences, Linköping University, Sweden; Andrea Koch, MD, Principal Investigator — Allergy Centre, University Hospital, Linköping, Sweden, Department of Pulmonary Medicine, University Hospital, Linköping, Sweden, and Department of Medical and Health Sciences, Linköping University, Sweden
Locations (13):
- Sweden (13):
  - Department of Pulmonary Medicine and Allergology, Sahlgrenska University Hospital, Gothenburg
  - Section of Pulmonary Medicine, Ryhov County Hospital, Jönköping
  - Section of Pulmonary Medicine and Allergology, County Hospital of Kalmar, Kalmar
  - Department of Pulmonary Medicine, University Hospital, Linköping
  - Department of Pulmonary Medicine and Allergy, Lund University Hospital, Lund
  - Section of Pulmonary Medicine, Malmö University Hospital, Malmo
  - Department of Pulmonary Medicine, Örebro University Hospital, Örebro
  - Department of Medicine, Skövde Hospital/KSS, Skövde
  - Department of Medicine, Trollhättan Hospital/NÄL, Trollhättan
  - Department of Medicine, Uddevalla Hospital, Uddevalla
  - Department of Pulmonary medicine, Umeå University Hospital, Umeå
  - Department of Pulmonary Medicine and Allergology, Uppsala University Hospital, Uppsala
  - Department of Medicine, Ystad Hospital, Ystad

REFERENCES:
- [Derived] Koch A, Bergman B, Holmberg E, Sederholm C, Ek L, Kosieradzki J, Lamberg K, Thaning L, Ydreborg SO, Sorenson S; Swedish Lung Cancer Study Group. Effect of celecoxib on survival in patients with advanced non-small cell lung cancer: a double blind randomised clinical phase III trial (CYCLUS study) by the Swedish Lung Cancer Study Group. Eur J Cancer. 2011 Jul;47(10):1546-55. doi: 10.1016/j.ejca.2011.03.035. Epub 2011 May 10. PMID 21565487